CLINICAL TRIAL: NCT04281732
Title: Visual Performance Measures in a Virtual Reality Environment for Assessing Clinical Trial Outcomes in Those With Severely Reduced Vision
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Sussex (Other)
Responsible Party: Principal Investigator, Ruth Hogg, Principal Investigator, Queen's University, Belfast
Other Study IDs: 17/NI/0002
Record Dates: First submitted 2019-08-12; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Low Vision; Retinitis Pigmentosa; Stargardt Disease 1; Stargardt Disease 3; Stargardt Disease 4; Albinism
Keywords: Virtual Reality; Quality of life
MeSH Terms: conditions — Vision, Low; Retinitis Pigmentosa; Stargardt Disease; Stargardt disease 3; Stargardt disease 4; Albinism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Virtual Reality Headset based tests — Visual task tests based on Oculus Rift

SUMMARY:
Purpose:

To validate a newly developed battery of performance-based tests of visual function to be presented using virtual reality. The tests are intended as potential outcome measures for clinical trials of treatments of eye disease: they measure visual performance in patients with low vision on visual tasks that a relevant for daily life.

DETAILED DESCRIPTION:
Aims of the Research Project:

1. To validate a new virtual reality (VR)-based battery of performance-based tests of visual function that are relevant for patients' daily lives.
2. To quantify the reproducibility of the performance-based tests.
3. To gather acceptability and ease-of-use data from patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants
2. Age 20-50
3. Bilateral sight impairment due to Stargardt's disease, retinitis pigmentosa or albinism.
4. Sight impairment criteria are as follows:

   * Visual acuity of 3 / 60 to 6 / 60 with a full field of vision.
   * Visual acuity of up to 6 / 24 with a moderate reduction of field of vision

Exclusion Criteria:

1. Any physical impairment that would make use of the virtual reality headset difficult or unsafe.
2. A history of vertigo or dizziness.

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients with Stargardt's disease, advanced retinitis pigmentosa and Albinism.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Test repeatability | All statistical analysis will take place once all data collection has ended, average 1 year.
  Bland and Altman analysis will be used to investigate the repeatability of the tests between visit 1 and visit 2.

SECONDARY OUTCOMES:
Ease of use and acceptability questionnaire | Responses from all participants will be collated and summarised at the end of the study, average 1 year.
  Modified from Tay et al, Br J Ophthalmol 2004;88:719-720
  Ask the following questions for virtual reality test:
  1. Was the test comfortable? If no- How?
  2. Was the test too long?
  3. How did you find the test? Would you describe it as easy or difficult? If you found it difficult- how?
  4. How would you feel if you knew you had to perform this test at every clinic appointment?
  5. Do you have any other comments about the test?

CONTACTS AND LOCATIONS:
Overall Officials: Ruth E Hogg, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- NI Clinical Research Facility, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT04281732/Prot_SAP_000.pdf